CLINICAL TRIAL: NCT03603782
Title: Ketone Plasma Kinetics After Oral Intake Of Different MCT Formulae
Brief Title: Ketone Plasma Kinetics After Oral Intake Of Different MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18.03.NRC
Record Dates: First submitted 2018-06-14; First posted 2018-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Proteins; Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 (Experimental)
  Interventions: Dietary Supplement: protein 5%; Dietary Supplement: protein 10%; Dietary Supplement: protein 15%; Dietary Supplement: B2: only breakfast (no product); Dietary Supplement: C2: 5% protein with breakfast; Dietary Supplement: D2: 5% protein 30 min before breakfast
- 2 (Experimental)
  Interventions: Dietary Supplement: 2.5% protein; Dietary Supplement: protein 10%; Dietary Supplement: protein 15%; Dietary Supplement: A2: Peptamen 1.5 Vanilla without Breakfast; Dietary Supplement: C2: 5% protein with breakfast; Dietary Supplement: D2: 5% protein 30 min before breakfast
- 3 (Experimental)
  Interventions: Dietary Supplement: 2.5% protein; Dietary Supplement: protein 5%; Dietary Supplement: protein 15%; Dietary Supplement: A2: Peptamen 1.5 Vanilla without Breakfast; Dietary Supplement: B2: only breakfast (no product); Dietary Supplement: D2: 5% protein 30 min before breakfast
- 4 (Experimental)
  Interventions: Dietary Supplement: 2.5% protein; Dietary Supplement: protein 5%; Dietary Supplement: protein 10%; Dietary Supplement: A2: Peptamen 1.5 Vanilla without Breakfast; Dietary Supplement: B2: only breakfast (no product); Dietary Supplement: C2: 5% protein with breakfast

INTERVENTIONS:
Dietary Supplement: 2.5% protein — 2.5%
  Arms: 2; 3; 4
Dietary Supplement: protein 5% — 5%
  Arms: 1; 3; 4
Dietary Supplement: protein 10% — 10%
  Arms: 1; 2; 4
Dietary Supplement: protein 15% — 15%
  Arms: 1; 2; 3
Dietary Supplement: A2: Peptamen 1.5 Vanilla without Breakfast — Peptamen withoug breakfast
  Arms: 2; 3; 4
Dietary Supplement: B2: only breakfast (no product) — only breakfast
  Arms: 1; 3; 4
Dietary Supplement: C2: 5% protein with breakfast — C2: 5% protein consumed with breakfast
  Arms: 1; 2; 4
Dietary Supplement: D2: 5% protein 30 min before breakfast — D2: 5% protein consumed 30 min before breakfast
  Arms: 1; 2; 3

SUMMARY:
This research project is aimed at identifying the MCT formulation matrixes that provide the highest ketoindex values and extended half-life, as well as to provide an initial evaluation of the GI tolerability of the various formula. For comparison, ketones salts and esters (food grade) will be also evaluated.

DETAILED DESCRIPTION:
Monocentric, open, randomized, controlled research project. The global research project will include several testing cycles as described in the figure 1. In each cycle, several research products (up to 4) will be tested on up to 20 participants in a partial or full cross-over design. Once cycle 1 is completed, blood parameters will be analysed and ketoindex will be calculated as area under the curve (AUC) of total ketones (BHB + AcA) over 4h / quantity of ingested MCTs in g. Based on ketoindex and ketones Thalf (T1/2: time to reach half of AUC-infinite of total ketones) values, new products will be developed for cycle 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50 years
2. Healthy men and women, based on the medical screening visit and medical history
3. BMI in the normal and overweight range 18.5 ≤ BMI ≤ 27.
4. Able to understand and to sign a written informed consent prior to study entry

Exclusion Criteria:

1. Any medication possibly impacting the postprandial glucose and insulin response (on anamnesis, to the opinion of the medical expert)
2. Any medication impacting dietary fat absorption and metabolism or impacting postprandial glucose and insulin response, to the opinion of the medical expert
3. Pregnancy (on anamnesis) and/or lactation
4. Known food allergy and food intolerance
5. Individuals undergoing either dietary or exercise mediated weight loss program prescribed by a health care professional
6. Individuals under ketogenic diets, or taking regular ketones products such as MCT, ketone esters or ketone salts (calcium, magnesium, sodium, potassium)
7. Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of bier
8. Having given blood within the last month, or willing to make a blood donation until one month following the end of the study
9. Participant having a hierarchical link with the research team members
10. Not expected to follow the protocol.
11. Smokers unable to stop for the day of the visit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
KetoIndex - plasma concentration | 4 hours
  KetoIndex calculated as area under the plasma concentration versus time curve (AUC) of total ketones (BHB + AcA) over 4 hours after MCT-based products consumption / quantity of ingested MCTs in gram.
total ketones (BHB+ACA) - Half-life time | 4 hours
  Half-Life time (T ½) calculated as time to reach half of Area under the plasma concentration versus time curve (AUC)-infinite of total ketones (BHB+ACA) after MCT-based products consumption.

SECONDARY OUTCOMES:
Ketones blood kinetic - Plasma concentration | 4 hours
  (Total Ketones, BHB, AcA) measured as plasma concentration versus time curve (AUCs) after MCT-based products consumption
Ketones blood kinetics - peak plasma concentration | 4 hours
  Peak Plasma Concentration (Cmax) of total Ketones, BHB, AcA MCT-based products consumption.
Ketones blood kinetics - time to maximum concentration | 4 hours
  Time to maximum concentration (Tmax) of total Ketones, BHB, AcA MCT-based products consumption.
Ketones blood kinetics - Half-life time | 4 hours
  Half-Life time (T ½) measured of total Ketones, BHB, AcA after MCT-based products consumption.
Medium chain fatty acid C8 and C10 - plasma concentration | 4 hours
  Measure of plasma concentration versus time curve (AUCs) of Medium chain fatty acid C8 and C10 after MCT-based products consumption
Medium chain fatty acid C8 and C10 - concentration | 4 hours
  Maximum plasma Concentration (Cmax) of Medium chain fatty acid C8 and C10 (and their metabolites) after MCT-based products consumption
Medium chain fatty acid C8 and C10 - Time to maximum concentration | 4 hours
  Time to maximum concentration (Tmax) of Medium chain fatty acid C8 and C10 (and their metabolites) after MCT-based products consumption
Medium chain fatty acid C8 and C10 - Half-life time | 4 hours
  Half-Life time (T ½) measured of Medium chain fatty acid C8 and C10 (and their metabolites) after MCT-based products consumption
Glucose and insulin - plasma concentration | 4 hours
  Measure of plasma concentration versus time curve (AUCs) of glucose and insuline after MCT-based products consumption
Glucose and insulin - peak plasma concentration | 4 hours
  Measure of maximum plasma concentration (Cmax) of glucose and insuline after MCT-based products consumption
Glucose and insulin - time to maximum concentration | 4 hours
  Measure of time to maximum concentration (Tmax) of glucose and insuline after MCT-based products consumption
Glucose and insulin- Half-life time | 4 hours
  Measure of Half-life time (T½) of of glucose and insuline after MCT-based products consumption
Gastro-intestinal tolerability assessment | 24 hours
  Gastro-intestinal tolerability assessment with visual analogue scales for each symptom of interest (i.e.) 1) Abdominal discomfort , 2) Decreased appetite, 3) Gastric reflux, 4) Nausea, 5) Diarrhea, 6) Headache). Each scale are from 0 (better outcome) to 100 (worst outcome).
Adverse event incidence | 24 hours
  Adverse events incidence

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, dr, Study Director — Nestec Ltd.
Locations (1):
- Metabolic Unit, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No